CLINICAL TRIAL: NCT05223387
Title: Tissue Level vs Bone Level Implants for Plural Restorations : a Multicentre Randomised Controlled Trial
Acronym: IBERICA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anthogyr (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1902
Record Dates: First submitted 2022-01-21; First posted 2022-02-04 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Dental Implants; Edentulous
Keywords: Anthogyr; dental; implant
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Anthogyr Axiom TL REG and corresponding Multi-Unit abutments
  Interventions: Device: Axiom TL REG
- Control Group (Active Comparator): Anthogyr Axiom BL REG and corresponding Multi-Unit abutment
  Interventions: Device: Axiom BL REG

INTERVENTIONS:
Device: Axiom TL REG — Anthogyr AXIOM TL Reg will be placed in healed bone crests in the mandible or maxilla for multiple teeth replacement, followed by a provisional prosthesis immediately loaded, if the patient needs a provisional.
  In each case, the MU abutment will be placed immediately after implant placement.
  Multi-Unit abutments are used to fix the prosthesis
  Other Names: Multi-Unit abutment
  Arms: Study Group
Device: Axiom BL REG — Axiom BL Reg implants will be placed in healed bone crests in the mandible or maxilla for multiple teeth replacement, followed by a provisional prosthesis immediately loaded, if the patient needs a provisional.
  In each case, the MU abutment will be placed immediately after implant placement.
  Multi-Unit abutments are used to fix the prosthesis
  Other Names: Multi-Unit abutment
  Arms: Control Group

SUMMARY:
Anthogyr Axiom Tissue-Level implants and corresponding Multi-Unit abutments recently enriched the available product range for dental surgeons. This Post-Market Clinical Follow-Up study aims at confirming the safety and performance of these products. The comparison with similar Anthogyr Axiom Bone-level implants will provide additional information on the effect of platform-switching in bone level maintenance for single and two-piece design at the implant level.

DETAILED DESCRIPTION:
This is a multicenter, comparative, prospective, randomized, controlled, post-market clinical follow-up (PMCF) study.

The total study duration for each patient should be 3 years. Anthogyr Axiom TL and BL REG and corresponding Multi-Unit abutments will be placed in healed bone crests in the mandible or maxilla for multiple teeth replacement, followed by a provisional prosthesis immediately loaded, if the patient needs a provisional.

In total 8 visits per patient are scheduled in this study

Implant and prosthesis survival, success, bone level changes, patient reported outcome, soft tissue assessment and adverse events (AEs) will be assessed.

The investigational devices are CE-(Conformité Européenne, meaning European Conformity) marked product.

3 centers will participate in Spain and Portugal.

The study and any amendments will be performed as far as possible according to International Organization for Standardization (ISO) 14155 and conform to the Declaration of Helsinki (last revision Fortaleza 2013) and local legal and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have voluntarily signed the Informed Consent Form before any study related procedures are performed, are willing and able to attend scheduled follow-up visits and agree that the pseudonymized data are collected and analyzed.
* Patients must be males or females who are a minimum of 18 years of age.
* Patients with a minimum of 4 weeks history of edentulism in the study area, in need of a multiple teeth replacement with dental implants
* Patients with complete soft tissue coverage of the socket at implant placement

Exclusion Criteria:

- Patients with inadequate bone volume and/or quality: Only minor and simultaneous bone augmentation procedures will be allowed where required for regeneration of minor defects. Insufficient bone volume and quality is defined as secondary exclusion criterion and the patient will be considered as screening failure.

* Uncontrolled systemic disease that would interfere with dental implant therapy (e.g. uncontrolled diabetes)
* Any contraindications for oral surgical procedures
* History of local irradiation therapy in the head / neck area
* Patients who are currently heavy smokers (defined >10 cigarettes per day or >1 cigar per day), or have ≥ 20 pack years who use chewing tobacco
* Medical conditions requiring chronic high dose steroid therapy or high dose anti-resorptive treatment
* Subjects who have undergone administration of any investigational device within 30 days of enrolment in the study
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance or unreliability
* Cognitive impairment that would interfere with the ability to perform adequate oral hygiene (assessed by Ottawa 3DY scale)
* Patients with chronic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2025-07-18 (Estimated); Study Completion 2027-07-18 (Estimated)

PRIMARY OUTCOMES:
Marginal Bone Level Change | 6 months,12 months, and 3 years after loading
  Change in crestal bone level measured by analysis of standardized peri-apical xrays [mm].

SECONDARY OUTCOMES:
Implant survival | 6 months,12 months, and 3 years after loading
  A surviving implant is an implant that is in place at the time of evaluation.
Prosthesis Survival | 6 months,12 months, and 3 years after prosthesis placement
  a surviving prosthesis is a prosthesis that is not broken at the time of evaluation.
14 item Oral Health Impact Profile (OHIP-14) | screening visit, 6, 12 months and 3 years after loading
  he local language version of the OPHIP-14 is a self-reported questionnaire that measures dysfunction, discomfort and disability attributed to oral conditions. The questionnaire focuses on seven dimensions of impact: Functional limitation; Pain; Psychological discomfort; Physical disability; Psychological disability; Social disability; Handicap. The patients will be asked to respond according to frequency of impact on a 5-point Likert scale coded never (score 0), hardly ever (score 1), occasionally (score 2), fairly often (score 3) and very often (score 4).

OTHER OUTCOMES:
Adverse Events | 3 years after inclusion
  Adverse Events will be recorded at every visit. Adverse Events will be recorded at every visit.
Device Deficiencies | 3 years after inclusion
  Adverse Events will be recorded at every visit. Any device complications and deficiencies will be recorded as Device Deficiencies.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Blanco Carrión, Pr.Dr., Principal Investigator — Universidad de Santiago de Compostela
Locations (3):
- Faculdade de Medicina Dentária da Universidade do Porto, Porto, Portugal
- Spain (2):
  - Universidad International de Catalunya, Barcelona
  - Universidad de Santiago de Compostela, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: No